CLINICAL TRIAL: NCT03665714
Title: Effects of Immunonutrition (Impact Oral®) in Patients Undergoing Surgery for Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17.01. CN. NHS
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-09

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impact Oral (Experimental): Preoperatively:
  1 bottle each time (250ml/bottle), 3 times per day, equivalent to approximately 1060.5kcal per day.
  Postoperatively:
  1. Patient should receive:
     * 1 bottle (250 ml each) per day of test product on D 1 and D 2 post surgery, corresponding to 353.5Kcal.
     * 2 bottles (250 ml each) per day of test product on D 3 and D 4 post surgery, corresponding to 707Kcal.
     * 3 bottles (250 ml each) per day of test product on D 5, D 6 and D 7 post surgery, corresponding to 1060.5 kcal.
  2. At the discretion of the authorized investigator/nutritionist, the amount of study products, can be increased to meet the daily caloric goal: 1500Kcal.
  Interventions: Other: Impact Oral; Other: Enteral Nutrition Emulsion(TPF-T)
- Enteral nutrition Emulsion(TPF-T) (Active Comparator): Preoperatively:
  272ml each time, 3 times per day, equivalent to approximately 1060.5kcal per day.
  Postoperatively:
  1. Patient should receive:
     * 272ml of control product on D 1 and D 2 post surgery, corresponding to 353.5Kcal.
     * 544ml of control product on D 3 and D 4 post surgery, corresponding to 707Kcal.
     * 816ml of control product on D 5, D 6 and D 7 post surgery, corresponding to 1060.5 kcal.
  2. At the discretion of the authorized investigator/nutritionist, the amount of study products, can be increased to meet the daily caloric goal: 1500Kcal.
  Interventions: Other: Impact Oral; Other: Enteral Nutrition Emulsion(TPF-T)

INTERVENTIONS:
Other: Impact Oral — Impact Oral belongs to Food for Special Medical Purpose (FSMP) according to China registration regulation, including Omega-3 fatty acids, Arginine and Nucleotides immunonutrition.
Other: Enteral Nutrition Emulsion(TPF-T) — TPF-T
  Other Names: Changnei Yingyang Ruji(TPF-T)

SUMMARY:
This study will evaluate the efficacy and safety of Impact Oral in Patients undergoing Surgery for Gastrointestinal Cancer, half of the participants will receive Impact Oral nutrition therapy, the other half will receive Enteral Nutrition Emulsion(TPF-T) therapy.

DETAILED DESCRIPTION:
The present protocol describes a randomized, active-controlled, open labelled study in which either IMPACT Oral or Enteral Nutrition Emulsion(TPF-T) will be given to surgical patients for 5 days before surgery and 7 days after surgery. Both of the study products include immunonutrition, but the nutrient proportion is different.

Prealbumin, C-reaction protein (CRP), Albumin，immunology parameters, the results of physical examination, vital signs, relevant nutrition- and safety-related laboratory parameters and the number, severity, seriousness, relatedness and outcome of Adverse Events (AEs) will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with upper or lower gastrointestinal cancer confirmed by histological method and scheduled for radical resection via open or laparoscopic surgery plus gastrointestinal reconstruction. Radiotherapy and/or Chemotherapy was not performed within 2 weeks before screening.
2. Age18-75 years old (include 18 and 75 years old).
3. Body Mass Index 18.5-28kg/m2 (include 18.5 and28kg/m2).
4. Life expectancy more than 3 months.
5. Plasma haemoglobin ≥ 90g/l.
6. Plasma albumin ≥2.5 g/dl.
7. No blood product infused within 1 week prior to screening.
8. Patients are informed for consent, and agreed to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Severe concomitant clinical conditions that could jeopardize the trial performance and follow-up.
2. Past history of gastrointestinal surgery or other treatment of digestive tract, and affect the nutrient absorption
3. Female patient who is pregnant or lactating woman.
4. Patient undergoing minor gastrointestinal cancer surgery such as confirmatory biopsy or endoscopy. Patient that has endoscopic tumour resection is also excluded.
5. Patient is not allowed any oral or enteral intake in the pre-operative phase of the study.
6. Having participated in another interventional clinical trial including those related to nutritional support within 4 weeks prior to the patient enrollment.
7. Other malignancies in the last 5 years (except for successfully treated in situ basocellular skin and in situ cervical uterine tumours).
8. Patient who is not willing and not able to comply with scheduled visits and the requirements of the study protocol.
9. Planned chemotherapy, radiotherapy or immunotherapy during the first 7 days following the surgical tumour resection.
10. Patient with liver and kidney dysfunction (alanine aminotransferase ALT ≥ 2 times the upper limit of normal; total bilirubin TBIL ≥ 2 times the upper limit of normal; creatinine Cr ≥ 2 times the upper limit of normal).
11. Known to have diabetes or fasting blood glucose≥ 10mmol/L.
12. Known to have hyperthreosis or hypothyreosis
13. Patient currently treated with Omega-3 fatty acid-containing fat emulsion, glutamine, thymosin, hormone, thyroxine, growth hormone, anti-TNF biological.
14. Known to have allergic history to any component of the investigational product.
15. Uncontrolled psychological disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change of Serum Prealbumin level | Change measures at baseline and Day 8 after surgery
  The change of serum prealbumin level on Day 8 after surgery compared with baseline (before study products treatment).

SECONDARY OUTCOMES:
Change of Serum Prealbumin level | Change measures at baseline and Day -1(before surgery) and Day1, Day3 after surgery
  Prealbumin at baseline and Day -1 before the day of surgery, and Day1 and Day 3 after the day of surgery.
Change of Albumin | Change measures at baseline, Day -1(before surgery),Day 1, 3, 8(after surgery)
  Albumin at baseline, Day-1 before the day of surgery, and on Day 1, 3 and 8 after the day of surgery.
Change of C-reactive protein | Change measures at baseline, Day -1(before surgery),Day1, 3, 8(after surgery)
  C-reactive protein at baseline, Day -1 before the day of surgery, and on Day 1, 3,8 after the day of surgery.
Change of Interleukin-6 (IL-6) | Change measures at baseline, Day -1(before surgery), Day 1, 3, 8(after surgery)
  Interleukin-6 (IL-6) at baseline, Day -1 before the day of surgery, and on Day1, 3 and 8 after the day of surgery
Change of CD4+/CD8+ | Change measures at baseline, Day -1(before surgery), Day1, 3, 8(after surgery)
  CD4+/CD8+ at baseline, Day-1 before the day of surgery, and on Day1, 3, 8 after the day of surgery(selected sites)
Incidence of postoperative Infections | up to Day 8 after surgery
  Incidence of postoperative infections up to Day 8 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianchun Yu, MD, Principal Investigator — Peiking Union Medical College Hospital; Gang Xiao, MD, Principal Investigator — Beijing Hospital; Yingjiang Ye, MD, Principal Investigator — Peiking University People's Hospital; Baogui Wang, MD, Principal Investigator — Tianjin Tumor Hospital
Locations (1):
- Peiking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No